CLINICAL TRIAL: NCT07287969
Title: Prospective Randomized Trial to Determine the Safety of Reusing Walking Boot Components for Patients Recovering From Acute Foot and Ankle Injuries
Brief Title: The Safety of Reusing Walking Boot Components for Patients Recovering From Acute Foot and Ankle Injuries
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Laura Bellaire, Principle Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 176418
Record Dates: First submitted 2025-12-14; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Foot Injuries; Ankle Injuries
Keywords: Reusing Walking Boot; PROCARE MaxTrax 2.0, Air, Tall; PROCARE MiniTrax; Safety
MeSH Terms: conditions — Foot Injuries; Ankle Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- New durable medical equipment (DME) walking boot (Active Comparator): A patient will be randomized to the "new" boot arm of the study.
  Interventions: Device: New durable medical equipment (DME) walking boot
- Re-used durable medical equipment (DME) walking boot (Experimental): A patient will be randomized to the "reuse" boot arm of the study.
  Interventions: Device: Re-used durable medical equipment (DME) walking boot

INTERVENTIONS:
Device: New durable medical equipment (DME) walking boot — The patient will be randomized and fitted with their designated DME boot.
  Other Names: PROCARE MaxTrax 2.0, Air, Tall; PROCARE MiniTrax
  Arms: New durable medical equipment (DME) walking boot
Device: Re-used durable medical equipment (DME) walking boot — The patient will be randomized and fitted with their designated DME boot.
  Other Names: PROCARE MaxTrax 2.0, Air, Tall; PROCARE MiniTrax
  Arms: Re-used durable medical equipment (DME) walking boot

SUMMARY:
The investigators primary purposes is to determine the safety of reusing a specific durable medical equipment (DME) item (walking boots) components for patients recovering from acute foot and ankle injuries.

The investigators secondary purpose is to determine the number of reuse episodes specific walking boot components can endure without increased failure rates.

To support further study of DME reuse, product design, and advocate for evolving regulations that promote waste reduction via development of reusable DME products in the US.

DETAILED DESCRIPTION:
The designation of an item as "durable medical equipment" (DME) implies the item is designed to be long-lasting and hold up to prolonged use. In practice, however, many DME items are utilized for a single patient after a single injury or procedure. This is particularly true in pediatric care, where patients are growing, and saving the item for later use is unlikely to maintain appropriate fit for the older child.

Walking boots, also termed CAM boots, are prescribed frequently in pediatric orthopaedic clinics across the country. These boots provide support, comfort, and immobilization while also allowing for removal to allow patients to begin wound care, range of motion exercises, and bathing. They provide a valuable transitional stage between casting and splinting and resumption of typical, unsupported ambulation and other activities. While differences in design exist between vendors, the vast majority of walking boots have a modular design including a base/sole attached to rigid medial and lateral posts, soft fabric/Velcro straps, and a soft cushioned liner. This modular design lends itself to opportunities for reuse and refurbishment, yet this is rarely considered.

Boots and other DME contribute considerable costs to patients and family. The costs of DME items vary widely, with simple items like canes costing less than $100 and custom items like power wheelchairs costing more than $5,000. In total, US spending on mobility-related DME items reached $1.5 billion in 2001, a figure that has likely grown exponentially over the past 2 decades due to inflation and supply chain shortages. Patients and health systems both encounter DME related charges, and health insurance payments for DME vary widely across payors. Provision of DME is a frequent cause of hospital discharge delays, contributing to lengthier hospital stays, prolonged immobilization, and greater cost of care. This is particularly true for low-income and uninsured families, perpetuating discrepancies in health equity and access to care. Charity care programs facilitate access to DME in some states, however Anti-Kickback statutes and other policies obstruct provision of free equipment in many systems.

Studies have shown that patients get little to no information related to appropriate reuse, recycling and other disposal programs for walking boots and other DME. Interview based studies suggest that equipment disposal options are simply not a part of discussions with patients-time with patients can be limited, time spent obtaining and fitting the DME item can be prolonged leaving little time to discuss other topics, and discussing disposal methods has been cited as sending a potential "mixed message" regarding the importance of the DME item itself.

Larger, more costly DME items owned by health systems including hospital beds and wheelchairs tend to be maintained by hospitals and care facilities so long as they can function without posing a threat to patient or staff safety. This is typically done through informal policies and guidance, borrowing from existing environmental service practices within a given facility for equipment cleaning and maintenance. Rental programs are available in many health systems for such items, with infrastructure to support their inspection, cleaning, and refurbishment as well as delivery and pick-up for some.

Hospitals that reuse DME see the double benefit of reduced budgets for purchasing new items and reduced costs of disposal-American health systems have been found to dispose of up to 10 billion dollars in equipment and supplies every year. Any fractional reduction in such practices would considerably reduce both cost and waste burden.

Smaller, patient-owned DME items, on the other hand, are not typically included in such reuse or rental programs. Instead, the majority of these items end up in landfills. They arrive in landfills either via residential or health system waste streams, depending on whether patients bring them back to their physician's office or leave them at home for a period before ultimately throwing them away. Some patients and clinics seek out alternative solutions including donation programs, parts salvage, recycling of core materials, and informally sharing the items with friends, family, and neighbors in need.

DME donation programs have emerged out of community charities, nonprofit organizations, and few health systems. Typically, specified items are collected informally from interested patients, then sent to low resource patients and communities in need without formalized or regulated inspection or reprocessing. Donation recipients can be local or represent communities abroad with partner organizations and/or medical mission programs. While generally well-intentioned, such programs beg the question-if reused DME items are good enough for these recipients, mustn't it also be good enough for everyone? "Why should someone who's poor get recycled equipment instead of new equipment" simply because they are impoverished?.

A further critical reason the medical community must reconsider the current practice of using of walking boots and other DME as single use items is related to waste. Attention to and scrutiny of the waste generated in and by health systems is growing, as is the recognition that orthopaedic surgeons and other healthcare practitioners have the ability to personally reduce the environmental harm caused by their practices. Like other waste reduction efforts, DME reuse programs should comprise part of hospital strategies to provide environmentally sustainable healthcare to communities.

While single use devices (SUDs) have seen a surge in popularity and adoption in the US, particularly with heightened concerns about contamination in the wake of the COVID pandemic, such items generate tremendous amounts of waste for which hospital systems are currently responsible.

Their increased utilization has also shifted hospital budgets and habits away from reusable items and bettering reprocessing pathways. There is a growing market for and interest in reprocessing SUDs and their components in the operating room setting, and regulations are shifting to support such efforts in the US and abroad. If physicians and their patients express interest in and willingness to utilize reuse programs, it is likely similar regulatory shifts will emerge to support such patterns in the realm of DME.

From an environmental stewardship standpoint, further study is needed surrounding optimal reuse pathways for walking boots and other DME. Life cycle assessments, which provide an estimate of the impact of specific products from cradle to grave, will inform opportunities to promote durability of reusable components and recycling or decomposition potential of those components (liners, straps) suited for only a single use. The sentiment, however, prevails that DME reuse and recycling represents the "right thing to do," and the only way to change routine behaviors is by reinforcing a sense of collective responsibility for the responsible and appropriate management of limited resources. Advancing research on the reuse potential of DME and other medical products is a necessary step in changing systems and organizational culture to promote the use of such items "for the duration of the lifespan for which they were built".

The DME specific boot the investigators use in the clinic is the PROCARE MaxTrax 2.0, Air, Tall or PROCARE MiniTrax depending on age and size of child.

ELIGIBILITY:
Inclusion Criteria:

* Patient is of ambulatory age
* Patient is ambulatory at baseline (i.e. prior to injury or intervention)
* Patient is recovering from an acute foot or ankle injury (bony or soft tissue)
* Patients expected to utilize the boot for <12 weeks total
* Prescribed in the outpatient clinic setting only

Exclusion Criteria:

* Patients with ongoing infection, skin lesions, or wounds
* Immunosuppressed patients
* Patients with autism or behavioral concerns
* Non ambulatory patients
* Fitted and provided in the operating room or inpatient settings

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Rate of skin based complications (%) | 1-2 weeks after boot receipt
  blisters, sores, erythema, rashes
Rate of skin based complications (%) | 4-weeks after boot receipt
  blisters, sores, erythema, rashes
Rate of skin based complications (%) | 3 months after boot receipt
  blisters, sores, erythema, rashes

CONTACTS AND LOCATIONS:
Overall Officials: Laura Bellaire, M.D., Principal Investigator — University of Utah Orthopaedics
Locations (1):
- University of Utah Orthopedics, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No